CLINICAL TRIAL: NCT06126861
Title: The Mass Balance Study of [14C]LP-168 in Chinese Healthy Subjects
Brief Title: The Mass Balance Study of LP-168 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN104
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Clinical Pharmacology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]LP-168 (Experimental): Using 14C-labeled LP-168 as a marker to investigate the absorption characteristic, as well as to evaluate the metabolism and elimination pathways in healthy subjects
  Interventions: Drug: [14C]LP-168

INTERVENTIONS:
Drug: [14C]LP-168 — single dose of 150 mg/100 μCi [14C] LP-168, orally suspension at fasted state

SUMMARY:
This study is a single-center, open-label, single-dose clinical pharmacokinetic study. The purpose of this study is to investigate the absorption characteristics, as well as to evaluate the metabolism and elimination pathways after a single oral dose of 150mg, 100μCi [14C]LP-168 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Aged 18-45 (including the boundary value);
* Body weight over 50 kg, the body mass index (BMI) is between 19 and 26 kg/m2 (including the boundary value);
* Subjects must sign the informed consent form voluntarily;
* Agree to abide the requirements of the study protocol, willing to communicate with the study doctor.

Exclusion Criteria:

* After a comprehensive physical examination, vital signs, laboratory tests and other examinations are abnormal and have clinical significance;
* Hepatitis B surface antigen or E antigen, hepatitis C virus antibody IgG (Anti-HCV IgG), human immunodeficiency virus antigen/antibody combined test (HIV-Ag/Ab) and Treponema pallidum antibody test positive;
* Subject with clinically significant abnormalities on ophthalmologic examination (slit lamp, intraocular pressure and fundus photography)
* Subject who have used any drug that inhibits or induces hepatic drug metabolizing enzymes or transporters during the screening period and within the previous 28 days;
* Subject who have taken any medication with inhibition gastric acid secretion during the screening period and within the previous 28 days
* Subject who have taken any anti-gastric acid medication during the screening period and within the previous 28 days
* Subject who have used any systemic medication during the screening period and within the previous 14 days
* Subject with a history of any clinically serious illness or disease or condition that, in the opinion of the investigator, may affect the results of the trial
* Subject with any condition that may affect the absorption of the drug
* Subject with history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, QT prolongation syndrome, or symptoms of QT prolongation syndrome or family history of these syndrome.
* Subject with major surgery during the screening period and within the previous 6 months or surgical incisions that have not fully healed
* Subject with allergies, such as a known history of allergy to two or more substances
* Subject with hemorrhoids or perianal disease with regular or ongoing blood in the stool, irritable bowel syndrome, inflammatory bowel disease
* Subject with habitual constipation or diarrhea
* Subject with alcohol abuse or regular use of alcohol in the 6 months prior to the screening period
* Subject with smoking >5 cigarettes per day before the first 3 months of the screening period
* Subject with drug abuse
* Subject who are subjected to long-term exposure to radioactive conditions
* Subject who have difficulty collecting blood or cannot tolerate venipuncture for blood collection
* Subject with participation in any other clinical trial during the screening period and within the previous 3 months
* Subject who have been vaccinated during the screening period and within the previous 1 month or who are scheduled to be vaccinated during the trial period
* Subject with plans to have children or donate sperm during the trial and within 1 year after completion of the trial
* Subject who had lost or donated up to 400 mL of blood during the screening period and within the previous 3 months, or those who had received a blood transfusion within 1 month;
* Subject with any factors that the investigator believes make participation in this trial inappropriate

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration of blood and plasma sample | Day 1- Day 8
  Use liquid scintillation counter to evaluate Radioactivity concentration of each sample
Radioactivity concentration of urine and feces sample | Day 1- Day 15
  Use liquid scintillation counter to evaluate Radioactivity concentration of each sample
Number of metabolites and its proportion in plasma, urine and feces. | Day 1- Day 15
  To study the metabolite profiling

SECONDARY OUTCOMES:
Plasma LP-168/Major Metabolic concentrations | Day 1- Day 8
  To determine the plasma concentrations of LP-168/Major Metabolic using LC-MS/MS.
Treatment emergent adverse events as assessed by CTCAE 5.0 | Day 1- Day 15
  To evaluate the safety after the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No